CLINICAL TRIAL: NCT07204938
Title: A Phase 3 Trial to Evaluate the Long-Term Safety and Efficacy of Navenibart in Participants With Hereditary Angioedema - ORBIT-EXPANSE
Brief Title: A Long-Term Study of Navenibart in Participants With Hereditary Angioedema
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Astria Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STAR-0215-302
Record Dates: First submitted 2025-09-30; First posted 2025-10-03 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: HAE; Angioedema; Long-Term; Safety
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema

STUDY DESIGN:
Intervention Model Description: In Part 1, adult participants who completed STAR-0215-301 and received navenibart will maintain their fixed dosing regimen from STAR-0215-301, whereas those who were randomized to placebo in STAR-0215-301 will receive navenibart 600 mg Q3M. In Part 2, adult participants may move among dosing regimens via the personalized dosing option (PDO) based on their individual needs. Adult participants who did not complete STAR-0215-301 may be eligible to enroll in Part 2 of STAR-0215-302 if they meet certain criteria. Adolescent participants will continue to receive their fixed dosing regimen from STAR-0215-301 until they turn 18 years of age.
Masking Description: All participants will knowingly receive navenibart, however participants, care providers, investigators, and outcome assessors will be blinded to their treatment arm for a duration specific to the individual.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Adult Dosing Regimen 1 (Experimental): Participants will receive 600 mg of navenibart every 3 months.
  Interventions: Drug: navenibart
- Adult Dosing Regimen 2 (Experimental): Participants will receive 300 mg of navenibart every 3 months.
  Interventions: Drug: navenibart
- Adult Dosing Regimen 3 (Experimental): Participants will receive 600 mg of navenibart every 6 months.
  Interventions: Drug: navenibart
- Adolescent Dosing Regimen 1 (Experimental): Participants will receive 300 mg of navenibart every 3 months.
  Interventions: Drug: navenibart

INTERVENTIONS:
Drug: navenibart — Navenibart will be administered as a subcutaneous injection.
  Other Names: STAR-0215

SUMMARY:
This is a Phase 3 multicenter trial in 2 parts to evaluate the long-term safety and efficacy of navenibart in adult and adolescent participants with hereditary angioedema (HAE) who participated in STAR-0215-301 (NCT06842823; ALPHA-ORBIT). Part 1 provides all participants with navenibart in a dose-controlled fashion; Part 2 introduces a personalized dosing option (PDO) for participants based on individual needs.

ELIGIBILITY:
Inclusion Criteria:

1. Participants from STAR-0215-301 who met one of the following conditions:

1. Completed STAR-0215-301 through the Day 181 visit
2. Withdrew from STAR-0215-301 but met the following criteria:

i. Received 2 doses of IP ii. completed ≥ 2 months of trial follow-up after the second dose of IP iii. Met other eligibility criteria as assessed by Investigator

Exclusion Criteria:

1. Participation in an investigational clinical trial other than STAR-0215- 301 in the 30 days or any exposure to an investigational drug (other than navenibart in STAR-0215-301) within 5 half-lives before informed consent/assent
2. Any exposure to angiotensin-converting enzyme (ACE) inhibitors or any estrogen containing medications with systemic absorption (such as hormonal contraceptives or hormone replacement therapy) within 30 days before Screening.
3. Known sensitivity to the ingredients in the formulation of IP

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Day 1 through Month 48

SECONDARY OUTCOMES:
Number of time-normalized investigator-confirmed HAE attacks | Day 1 through Month 48
Number of moderate or severe investigator-confirmed HAE attacks | Day 1 through Month 48
Number of investigator-confirmed HAE attacks that require on-demand treatment | Day 1 through Month 48
Percent reduction in monthly investigator-confirmed HAE attacks | Day 1 through Month 48
Time to first investigator-confirmed HAE attack after first dose | Day 1 through Month 48
The number of participants responding to treatment, defined as a ≥ 50%, ≥ 70%, or ≥ 90% reduction in investigator-confirmed HAE attack rate | Day 1 through Month 48
Number of participants with no investigator-confirmed HAE attacks | Day 1 through Month 48
Angioedema Quality of Life questionnaire total score | Day 1 through Month 48
  The Angioedema Quality of Life Questionnaire (AE-QoL) consists of 17 questions divided into four domains: functioning (4 questions), fatigue/mood (5), fears/shame (6), and food/nutrition (2). Each question is answered on a 5-point scale from "never" to "very often." Scores are calculated for each domain and then normalized to a scale from 0 to 100, where 0 represents the best possible quality of life and 100 the worst.

CONTACTS AND LOCATIONS:
Locations (1):
- Site 2, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No